CLINICAL TRIAL: NCT07243600
Title: Improving Neurological Health With Acetylcholine Via Neuroplasticity-based Computerized Exercise in Mild Cognitive Impairment (INHANCE-MCI)
Brief Title: Improving Neurological Health With Acetylcholine Via Neuroplasticity-based Computerized Exercise in Mild Cognitive Impairment
Acronym: INHANCE-MCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSC-0703-25
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speed Training (Experimental): Computerized speed-based cognitive training requiring a total maximum of 70 treatment sessions, up to 7 sessions per week, 30 minutes per session.
  Interventions: Other: Computerized speed-based cognitive training
- Executive Function Training (Active Comparator): Computerized executive function cognitive training requiring a total maximum of 70 treatment sessions, up to 7 sessions per week, 30 minutes per session.
  Interventions: Other: Computerized executive function cognitive training

INTERVENTIONS:
Other: Computerized speed-based cognitive training — Thirty minutes of training on computerized exercises that targets visual processing speed, memory, attention and alertness.
  Arms: Speed Training
Other: Computerized executive function cognitive training — Thirty minutes of training on computerized exercises that target executive function.
  Arms: Executive Function Training

SUMMARY:
This study is a validation study to evaluate efficacy of two neuroplasticity-based, computerized cognitive training programs to improve neurological and neuropsychological health in older adults with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate will evaluate the impact of speed training to change cholinergic signaling, cognitive performance, and functional abilities in patients with MCI, as evidenced by [18F]fluoroethoxybenzovesamicol (FEOBV) positron-emission tomography (PET) and standard measures of cognition and function.

The investigators will employ a prospective, double-blind, parallel-arm, active-controlled, randomized clinical trial in patients with clinically-defined mild cognitive impairment aged 65 and above with a baseline MoCA of 18-26 inclusive.

Approximately 84 participants will be consented to ensure the successful completion of at least 70 participants (post 20% attrition). Participants will then complete the Screening (V0) assessments to determine eligibility. Following inclusion, participants will complete the Baseline (V1) assessments, PET imaging and structural MRI scan; participants will then be randomized into either the speed-based brain training or an active control of visual non-speeded computerized games and will engage in approximately 35 hours of program use for the 10-week Intervention Period. Following the 10-week intervention, participants will complete a Post-Intervention (V2) assessment, and PET imaging to evaluate changes in cognitive function. Participants will then stop using their assigned program for 3 months and return for a Follow-up (V3) end-of-study assessment and PET imaging to evaluate the endurance of changes in cognition, function, and behavior in the absence of further program use.

ELIGIBILITY:
Inclusion Criteria:

1. Potential participant must be 65 years or older at the time of study screening.
2. Potential participant must have MCI as defined by:

   * Total score between 18-26 inclusive on the Montreal Cognitive Assessment (MoCA)
   * Cognitive concern by participant, informant, or clinician and evidence of preserved functional abilities as defined as a Clinical Dementia Rating (CDR) of 0.5 with a memory score of 0.5 or 1.
3. Potential participant must have a study partner/informant defined as any acquaintance (e.g., family member, friend, neighbor, clinician) who has regular (at least monthly) interactions (in person or remote) with the participant.
4. If potential participant reports use of medications typically prescribed for dementia such as, but not limited to, Namenda, Memantine, Namzaric, Donepezil, Aricept, Rivastigmine, Exelon, Razadyne, Galantamine, Reminyl, Aducanumab, Leqembi or Lecanemab, Donanemab, the dose must be stable for at least 12 weeks prior to study enrollment.
5. Potential participant must demonstrate adequate decisional capacity, in the judgment of the investigator, and capable of to making an informed decision regarding their participation in this research study.
6. Potential participant must be likely able to complete all study activities and outcome measures in the judgment of the investigator.
7. Potential participant must have the visual, auditory, and motors capacity to use the computerized intervention in the judgment of the investigator.
8. Potential participant must be able to communicate in either English or French.

Exclusion Criteria:

1. Potential participant has an existing diagnosis of major neurocognitive disorder at screening (DSM-IV).
2. Potential participant who answered 'yes' to question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the C-SSRS or 'yes' to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the C-SSRS "Suicidal Behavior" if the ideation or behavior occurred within 2 months from Participant's date of consent (as recommended by the FDA for treatment trials.)
3. Potential participant scores >10 on the Geriatric Depression Scale - Short Form (GDS-SF).
4. Potential participant has previously completed 10 or more hours of the computerized cognitive intervention program manufactured by Posit Science.
5. Potential participant is participating in a concurrent clinical trial (involving an investigational pharmaceutical, behavioral treatment, medical device or other) that, in the judgment of the investigator, could affect the outcome of this study.
6. Potential participant is pregnant or breastfeeding.
7. Potential participant has claustrophobia or implantation with any medical devices above the waist that may concentrate radio frequency fields or have other medical issues that may frustrate participation in MRI/PET imaging procedures.
8. Potential participant has a history of large vessel stroke with significant residual motor or cognitive impairment.
9. Potential participant has a history of moderate to severe traumatic brain injury with residual cognitive symptoms.
10. Potential participant has a history of brain tumor.
11. Potential participant has a congestive heart failure diagnosis.
12. Potential participant has a primary diagnosis of idiopathic Parkinson's disease.
13. Potential participant has multiple sclerosis or Amyotrophic lateral sclerosis diagnosis.
14. Potential participant has evidence of a non-neurodegenerative neurological disorder that would interfere with the ability to carry out study activities.
15. Potential participant has has evidence of any other unstable medical conditions that would interfere with the ability to carry out study activities or cause fluctuations in cognition (for example, but not limited to, unstable diabetes, chronic obstructive pulmonary disorder dependent on oxygen).
16. Potential participant has any other clinically significant or unstable medical condition (for example, but not limited to, ongoing alcohol dependency or drug abuse, schizophrenia, psychosis) that in the investigator's opinion would interfere with the ability to carry out study activities.
17. Potential participant is undergoing or plans to undergo surgery requiring anesthesia, chemotherapy, or radiation treatment in the six months following screening (can be rescreened and enrolled later).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-03-03 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Global cholinergic signaling using [18F]fluoroethoxybenzovesamicol (FEOBV) positron-emission tomography (PET) | at 3 months (post-intervention)
  FEOBV standard uptake value ratios (SUVR) in the global cortex ROI. Higher score is better.

OTHER OUTCOMES:
Change in Memory-based cholinergic signaling in hippocampus gyrus using [18F]fluoroethoxybenzovesamicol (FEOBV) positron-emission tomography (PET) | at 3 months (post-intervention)
  FEOBV-PET standard uptake value ratios (SUVR) hippocampus gyrus using Matched MNI-space region via Hammers Atlas. Higher score is better.
Change in Memory-based cholinergic signaling in parahippocampal gyrus using [18F]fluoroethoxybenzovesamicol (FEOBV) positron-emission tomography (PET) | at 3 months (post-intervention)
  FEOBV-PET standard uptake value ratios (SUVR) parahippocampal gyrus using Matched MNI-space region via Hammers Atlas. Higher score is better
Change in NIH EXAMINER Executive Composite Score | at 3 months (post-intervention) and at 6 months (follow-up)
  The NIH EXAMINER is a computer based battery of executive function tests which yields a total or 'composite' score to represent global executive functioning. Higher score is better.
Change in Clinical Dementia Rating Sum of Boxes (CDR-SB) Score | at 3 months (post-intervention) and at 6 months (follow-up)
  The Clinical Dementia Rating (CDR) Scale is a validated assessment for evaluating severity of dementia. Lower score is better.
Change in Double Decision train-to-task Assessment Score | at 3 months (post-intervention) and at 6 months (follow-up)
  This is a computerized assessment that serves as a positive control for task learning. A single exposure duration (in milliseconds) required for users to achieve approximately 80% criterion accuracy in identification of central and peripheral targets. Higher score is better.
Change in Eye-tracking Test | at 3 months (post-intervention) and at 6 months (follow-up)
  Eye movements will be measured to determine acetylcholinergic function over time. A series of oculomotor tasks will be presented sequentially on an iPad Pro for approximately 20 minutes. Each task consists of visual stimuli designed to elicit specific eye movements. The iPad's front-facing camera will record facial and eye movements during task performance.

CONTACTS AND LOCATIONS:
Overall Officials: Mouna Attarha, PhD, Principal Investigator — Posit Science Corporation